CLINICAL TRIAL: NCT02198209
Title: Liraglutide Actions on the Liver: Effects on Glucose Phosphorylation
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator decided not to move forward with study prior to study start date
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Marilyn Ader, PhD, Associate Director, Diabetes & Obesity Research Institute, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: U1111-1138-7223
Record Dates: First submitted 2014-07-21; First posted 2014-07-23 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Type 2 Diabetes
Keywords: liraglutide; GLP-1; liver glucokinase
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Maturity-Onset Diabetes of the Young, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- single arm (Other): Liraglutide (Victoza)
  1. acute study: one injection of 0.6 mg s.c. before IVGTT
  2. chronic study: 6 weeks of daily liraglutide administration (1 week at 0.6 mg, 1 week at 1.2 mg, 4 weeks at 1.8 mg, s.c).
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide — 1. acute study: one injection of 0.6 mg s.c. before IVGTT
  2. chronic study: 6 weeks of daily liraglutide administration (1 week at 0.6 mg, 1 week at 1.2 mg, 4 weeks at 1.8 mg, s.c).
  Other Names: Victoza

SUMMARY:
Type 2 diabetes is a chronic disease that has reached epidemic proportions. In order to improve our strategies for preventing and treating type 2 diabetes the investigators need to better understand the mechanism of this disease, and the way in which current therapies, such as the drug liraglutide, work to control blood sugar. It is known that liraglutide acts via increasing the secretion of the hormone insulin from the pancreas, hormone that in turn controls blood sugar. However, it is not known whether liraglutide also has actions on the liver. Animal studies have suggested that liraglutide might act by controlling the liver enzyme glucokinase (GCK), an enzyme that increases blood sugar uptake by the liver. This could be a crucial mechanism in which liraglutide controls blood sugar independently of insulin, thus making it beneficial not only in type 2 but also in type 1 diabetes. The effect of liraglutide on GCK activity has not been yet measured in humans. The investigators propose to investigate the acute and chronic effect of liraglutide on GCK by using a simple, widely used procedure (an IntraVenous Glucose Tolerance Test-IVGTT) and a novel approach (mathematical modeling of data obtained from this procedure), to assess GCK activity in people with type 2 diabetes. The investigators will first compare data obtained form 2 IVGTTs (with and without liraglutide) performed 1 week apart (acute effect). The investigators will then give liraglutide to patients for 6 weeks and do another IVGTT to measure GCK activity (chronic effects). Data obtained from this study will be used to further understand the mechanism of liraglutide action and how to better employ our current therapeutic options and develop new strategies for preventing and treating diabetes.

DETAILED DESCRIPTION:
It is known that liraglutide impacts favorably glucose homeostasis in type 2 diabetic patients, but not the exact mechanism of this effect. In particular, liraglutide's acute and chronic effects on the liver are not well understood. The aim of our study is to determine whether liraglutide acutely and/or chronically changes hepatic GCK activity in vivo in type 2 diabetic patients, and to quantify this effect. We hypothesize that liraglutide increases GCK activity and that this results in increased hepatic glucose uptake, contributing to a lowering of glycemia.

Our specific aims are:

1. to measure liraglutide's acute effect on GCK activity changes in vivo in type 2 diabetic patients;
2. to assess whether chronic treatment with liraglutide determines a change in liver GCK activity in type 2 diabetic patients, as assessed during an IVGTT.

We expect that liraglutide acutely and/or chronically increases GCK activity, thus contributing to higher liver glucose uptake and lower glycemia.

Primary endpoints

1. GCK activity (acute effect) during IVGTTs with and without liraglutide administration. GCK activity will be calculated based on lactate and glucose measurements during the IVGTT
2. GCK activity during IVGTTs before and after 6 weeks of liraglutide treatment (IVGTT3).

Secondary endpoints

1. SI-IVGTT (insulin sensitivity during an intravenous glucose tolerance test) as quantified by the MINMOD analysis of the IVGTT
2. Acute insulin response to glucose (AIRg) and the disposition index (DI-MINMOD), the ability of beta cell to compensate for changes in insulin sensitivity.

This is a study designed to investigate the effect of liraglutide in type 2 diabetes therefore subjects are selected from type 2 diabetes population of the Los Angeles basin area. The study population is represented by type 2 diabetics (age 18-65 y old, T2DM diagnosed by current American Diabetes Association diagnostic criteria ( HbA1c ≥ 6.5 % or fasting plasma glucose ≥ 126 mg/dl or 2h plasma glucose ≥ 200 mg/dL during an OGTT or in a patient with classic symptoms of hyperglycemia or hyperglycemic crisis a random plasma glucose ≥ 200 mg/dl).

ELIGIBILITY:
Inclusion Criteria:

* 18- 65 years of age (inclusive)
* Ability to provide informed consent before any trial-related activities
* Ability to communicate effectively with research staff
* Ability to return for follow up visit
* Adequate IV access
* If a female of childbearing potential, non-pregnant and taking reliable contraception
* Documented T2DM (per most recent American Diabetes Association criteria);
* Drug naïve or treated with metformin only;
* Diabetes should be well controlled (as defined by HbA1 ≤ 7.5%, FPG <180 mg/dl).

Exclusion Criteria:

* Pregnant, breast-feeding or the intention of becoming pregnant or not using adequate contraceptive measures
* Presence of cancer or any clinically significant cardiac, respiratory, renal, hepatic, gastrointestinal, endocrinological, haematological, neurological, or psychiatric diseases or disorders (inclusion will be discussed with attending physician)
* Liver disease; history of alcoholism.
* Known or suspected allergy to liraglutide
* Contraindications to liraglutide: patients with a personal or family history of medullary thyroid carcinoma or in patients with Multiple Endocrine Neoplasia syndrome type 2
* Patients with a history of pancreatitits
* Patients that have been treated with drugs that promote weight loss (e.g., Xenical® [orlistat], Meridia® [sibutramine], Acomplia® [rimonabant], Acutrim® [phenylpropanolamine], or similar over-the-counter medications) within 3 months of study start
* Patients that have been treated with diabetes drugs: injectables, (e.g GLP-1R agonists (Byetta® [exenatide], Victoza® [liraglutide]) amylin analogues; insulin and insulin analogues) or oral agents other than metformin (e.g.DPP-IV- inhibitors (Januvia® [sitagliptin], Onglyza® [saxagliptin] or Janumet® [sitagliptin and metformin]),insulin sensitizers (thiazolidindiones: pioglitazone [Actos®]); or sulfonylureas) within 3 months of study start.
* The receipt of any investigational drug within 3 months prior to study start.
* Type 1 diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Liver glucokinase activity (acute effect) | 12 months
  We will measure liver glucokinase (GCK) activity 'in vivo' during IVGTTs with and without liraglutide administration
Liver glucokinase activity (chronic effect) | 12 months
  We will measure liver glucokinase (GCK) activity 'in vivo' during IVGTTs before and after 6 weeks of daily liraglutide administration

SECONDARY OUTCOMES:
insulin sensitivity | 12 months
  We will measure SI-IVGTT (insulin sensitivity during an intravenous glucose tolerance test) as quantified by the MINMOD analysis of the IVGTT.
Acute insulin response to glucose and the disposition index | 12 months
  We will assess the acute insulin response to glucose (AIRg) and the disposition index (DI-MINMOD)(the ability of beta cell to compensate for changes in insulin sensitivity)

CONTACTS AND LOCATIONS:
Overall Officials: Viorica Ionut, MD PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States